CLINICAL TRIAL: NCT05843461
Title: The Pulmonary Index of Microcirculatory Resistance: a Novel Hemodynamic Index for Invasively Assessing the Pulmonary Vasculature
Brief Title: PIMR and Pulmonary Vascular Disease
Status: Completed | Type: Observational
Sponsor: University of California, Los Angeles (Other)
Collaborators: Abbott (Industry)
Responsible Party: Principal Investigator, Rushi V. Parikh, Principal Investigator, University of California, Los Angeles
Other Study IDs: IRB#22-001643
Record Dates: First submitted 2023-04-24; First posted 2023-05-06 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Pulmonary Hypertension
Keywords: Pulmonary Hypertension; Pulmonary Arterial Hypertension; Index of Microcirculatory Resistance; Chronic Thromboembolic Disease; Pulmonary Index of Microcirculatory Resistance
MeSH Terms: conditions — Hypertension, Pulmonary; Pulmonary Arterial Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Controls: 10 patients without pulmonary hypertension (mean PA pressure less than 20 mmHg on RHC)
  Interventions: Other: Pulmonary Index of Microcirculatory Resistance
- PAH: 10 patients with PAH
  Interventions: Other: Pulmonary Index of Microcirculatory Resistance; Other: Right Ventricle Index of Microcirculatory Resistance; Other: Pulmonary artery OCT
- CTEPH: 10 patients with CTEPH
  Interventions: Other: Pulmonary Index of Microcirculatory Resistance; Other: Right Ventricle Index of Microcirculatory Resistance; Other: Pulmonary artery OCT

INTERVENTIONS:
Other: Pulmonary Index of Microcirculatory Resistance — PIMR measurement involves placing a coronary pressure wire in the pulmonary arteries and making pressure/time measurements during maximal flow down the artery. PIMR of the right and left pulmonary arteries will be obtained.
  Other Names: PIMR
Other: Right Ventricle Index of Microcirculatory Resistance — RV-IMR measurement involves placing a coronary pressure wire in the acute marginal branch of the right coronary artery and making pressure/time measurements during maximal flow down the artery.
  Other Names: RV-IMR
  Groups: CTEPH; PAH
Other: Pulmonary artery OCT — OCT of the pulmonary artery involves advancing an OCT catheter over the pressure wire to image the pulmonary artery. OCT of the right and left pulmonary arteries will be performed.
  Groups: CTEPH; PAH

SUMMARY:
The findings from this innovative, first-in-man, prospective pilot study will elucidate the role of PIMR and RV-IMR in pre-capillary PH. The study cohort will consist of patients with pulmonary pressures ranging from normal (advanced lung disease patients undergoing lung transplant evaluation) to severe PH (PAH and CTEPH patients), and thus will allow for identification of a PIMR cutoff. Participants will include: 1) advanced lung disease patients undergoing bilateral heart catheterization as part of their pre-lung transplant work-up, and 2) newly referred patients to PAH and CTEPH clinics undergoing bilateral heart catheterization as part of standard of care work-up. All participants will undergo PIMR testing, and those with pre-capillary PH will also undergo pulmonary OCT and measurement of RV-IMR. The study seeks to define the relationship between PIMR and PH and to establish the PIMR threshold that identifies pulmonary microvascular dysfunction as well as to evaluate the association of PIMR and pulmonary vascular remodeling on OCT in patients with pre-capillary PH. In addition, the study will assess the relationship between RV-IMR and RV pressure overload among patients with pre-capillary PH.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old
* Able to provide informed written consent.
* Patients with 1) advanced lung disease requiring standard-of-care bilateral heart catheterization as part of lung transplant evaluation in whom mPAP < 20 mmHg on RHC, or 2) PAH/CTEPH (i.e. pre-capillary PH) undergoing standard-of-care bilateral heart catheterization as part of their work-up/treatment

Exclusion Criteria:

* Contraindicated to undergo fluoroscopy and/or coronary angiography (e.g. pregnancy)
* Chronic kidney disease (serum creatinine ≥ 2.0 mg/dL)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled to undergo standard-of-care right and left heart catheterization either for evaluation of suspected or known pulmonary hypertension (PAH or CTEPH) or for lung transplant evaluation in the setting of advanced lung disease
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2023-01-10 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Pulmonary Index of Microcirculatory Resistance (PIMR) | Baseline
  PressureWire advanced to distal third of segmental pulmonary artery (PA) for measurement of pulmonary hemodynamics. The derivation of IMR involves the application of Ohm's law (V=IR) to the coronary microcirculatory circuit, where the relationship between resistance (R) = IMR, voltage (V) = pressure (P), and current (I) = flow (Q) can be expressed as follows: IMR = ∆P/Q. ∆P = the change in pressure across the microvasculature (mean distal coronary artery pressure [Pd] - coronary venous pressure (Pv); Pv is typically disregarded because it is negligible relative to Pd. Based on the principles of thermodilution, flow is inversely proportion to mean transit time (Q ~ 1/Tmn). Lastly, the minimal achievable resistance occurs during maximal hyperemic flow when all available microvessels have theoretically been recruited. Hence, the calculation of IMR simplifies to the following formula: IMR = Pd (pulmonary artery) x TmnHyp.
Right Ventricle Index of Microcirculatory Resistance (RV-IMR) | Baseline
  PressureWire advanced to distal third of acute marginal branch of the right coronary artery (RCA) for measurement of pulmonary hemodynamics. The derivation of IMR involves the application of Ohm's law (V=IR) to the coronary microcirculatory circuit, where the relationship between resistance (R) = IMR, voltage (V) = pressure (P), and current (I) = flow (Q) can be expressed as follows: IMR = ∆P/Q. ∆P = the change in pressure across the microvasculature (mean distal coronary artery pressure [Pd] - coronary venous pressure (Pv); Pv is typically disregarded because it is negligible relative to Pd. Based on the principles of thermodilution, flow is inversely proportion to mean transit time (Q ~ 1/Tmn). Lastly, the minimal achievable resistance occurs during maximal hyperemic flow when all available microvessels have theoretically been recruited. Hence, the calculation of IMR simplifies to the following formula: IMR = Pd (RCA marginal branch) x TmnHyp.
OCT-derived pulmonary artery wall thickness | Baseline
  A Dragonfly Optis OCT catheter (Abbott) will be advanced over the PressureWireX to the distal left lower lobe segmental pulmonary artery (luminal diameter < 5 mm and minimal length of 50 mm). OCT images of the pulmonary artery will be recorded via automatic pullback and analyzed offline in a blinded manner.
OCT-derived thickness-diameter ratio | Baseline
  A Dragonfly Optis OCT catheter (Abbott) will be advanced over the PressureWireX to the distal left lower lobe segmental pulmonary artery (luminal diameter < 5 mm and minimal length of 50 mm). OCT images of the pulmonary artery will be recorded via automatic pullback and analyzed offline in a blinded manner.
OCT-derived wall-area ratio | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Rushi Parikh, MD, Principal Investigator — University of California, Los Angeles
Locations (1):
- Ronald Reagan UCLA Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No